CLINICAL TRIAL: NCT00489957
Title: Speckle Tracking and Function Assessment in Pediatric Patients
Brief Title: Speckle Tracking in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Full Professor, Emory University
Other Study IDs: IRB00001930
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Cardiomyopathy
Keywords: congenital cardiac disorders; echocardiography
MeSH Terms: conditions — Cardiomyopathies; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normals
- Cardiomyopathy

SUMMARY:
An echocardiogram, also called a cardiac ultrasound or echo, is a medical test that takes pictures of the heart using sound waves. It shows images of the structures of the heart without using radiation. During the last year, the FDA has approved a new technology called Speckle Tracking that can look at the heart wall motion and contraction (pumping or squeezing) abnormalities. The study will also employ tissue Doppler and 3-Dimensional echo and uses the same echocardiographic machines which are used right now. The machines are upgraded with the new software application. This new technology is currently being used in adults, but unfortunately, there is almost no published data about normal heart function in infants and children using this technology. It is known from other technologies that the developing child's heart is not the same as an adult.

The investigators wish to study this new technology and compare it to other technologies currently being used.

DETAILED DESCRIPTION:
This study will be done primarily by software analysis.

The investigators wish to enroll a total of 70 patients aged newborn to 17 years old. The patients will be divided into three groups: (1) 0-2 years (2) 2-10 years (3) 10-17 years of age. 59 of the patients will be normal volunteers - siblings of patients receiving routine echoes or siblings of patient caregivers at Children's Healthcare of Atlanta. The investigators will age-match those patients with twenty patients with known or suspected heart muscle dysfunction (not working properly) already scheduled for a routine echo. For the patients scheduled for a routine echo, the patient and parent/guardian will be approached prior to the routine echo being performed. If they consent/assent, it will take an additional 10-15 minutes to obtain the research images after their routine images have been obtained. The healthy volunteers will be screened from the siblings of the patients receiving a routine echo or from siblings of patient caregivers, the study explained and informed consent/assent obtained. It will take approximately 30 minutes to obtain the research images.

By studying this new technology, the investigators will be able to find out whether it will be able to give us useful information on how the heart muscle contracts, the coordination of these contractions and if it may indicate new areas for treatment.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers

* No known heart disease
* Age of birth to 17 years.
* Patients will be compared to age appropriate controls.
* Stable clinical condition
* Able and willing to sign informed assent (where appropriate) and consent

Study Group

* Suspected or known heart muscle dysfunction or cardiomyopathy.
* Age of birth to 17 years
* Stable clinical condition
* Able and willing to sign informed assent (where appropriate) and consent

Exclusion Criteria:

* Patients who do not have structurally normal left ventricles, have unstable or irregular heart rhythms.
* Patients not in stable clinical condition
* Unable or unwilling to sign informed consent and/or assent.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborn - 17 year old patients at Children's Healthcare of Atlanta Egleston campus with known or suspected heart muscle dysfunction already scheduled for a routine echo. Also looking at normal controls.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The investigators wish to study a new technology called Speckle Tracking and compare it to other technologies currently being used. | Retrospective Chart Review
  An echocardiogram, also called a cardiac ultrasound or echo, is a medical test that takes pictures of the heart using sound waves. It shows images of the structures of the heart without using radiation. During the last year, the FDA has approved a new technology called Speckle Tracking that can look at the heart wall motion and contraction (pumping or squeezing) abnormalities. The study will also employ tissue Doppler and 3-Dimensional echo and uses the same echocardiographic machines which are used right now. The machines are upgraded with the new software application. This new technology is currently being used in adults, but unfortunately, there is almost no published data about normal heart function in infants and children using this technology. It is known from other technologies that the developing child's heart is not the same as an adult.
  The investigators wish to study this new technology and compare it to other technologies currently being used.

CONTACTS AND LOCATIONS:
Overall Officials: Derek A Fyfe, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States